CLINICAL TRIAL: NCT02768337
Title: Cambridge Brain Mets Trial 1: A Proof-of-principle Phase 1b/Randomised Phase 2 Study of Afatinib Penetration Into Cerebral Metastases for Patients Undergoing Neurosurgical Resection, Both With and Without Prior Low-dose, Targeted Radiotherapy
Brief Title: Cambridge Brain Mets Trial 1
Acronym: CamBMT1
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Slow recruitment
Sponsor: Cambridge University Hospitals NHS Foundation Trust (Other)
Collaborators: Boehringer Ingelheim (Industry); Cancer Research UK (Other); University of Cambridge (Other); The Brain Tumour Charity (Other)
Responsible Party: Principal Investigator, Richard D. Baird MD PhD, Dr Richard Baird, Cambridge University Hospitals NHS Foundation Trust
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: CamBMT1; 2013-002398-23 (EudraCT Number); 1200.206 (Other Grant/Funding Number: Boehringer-Ingelheim); 146009 (Other: IRAS)
Record Dates: First submitted 2016-04-28; First posted 2016-05-11 (Estimated); Last update posted 2024-01-31 (Actual); Status verified 2024-01

CONDITIONS: Lung Cancer; Breast Cancer; Brain Cancer; Advanced Breast Cancer; Advanced Lung Cancer
Keywords: brain metastasis; operable brain metastasis
MeSH Terms: conditions — Lung Neoplasms; Breast Neoplasms; Brain Neoplasms | interventions — Afatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Arm 1: Afatinib only at Recommended Phase 2 dose (RP2D) (Other): No targeted radiotherapy. Afatinib at Recommended Phase 2 Dose for 11 days.
  Interventions: Drug: Afatinib
- Arm 2: Afatinib RP2D + 2 Gy targeted radiotherapy (Experimental): Patient will receive the RP2D of afatinib for 11 days and will receive targeted radiotherapy at a dose level of 2 Gy on Day 10 of treatment.
  Interventions: Drug: Afatinib; Radiation: 2 Gy targeted radiotherapy
- Arm 3: Afatinib RP2D + 4 Gy targeted radiotherapy (Experimental): Patient will receive the RP2D of afatinib for 11 days and will receive targeted radiotherapy at a dose level of 4 Gy on Day 10 of treatment.
  Interventions: Drug: Afatinib; Radiation: 4 Gy targeted radiotherapy

INTERVENTIONS:
Drug: Afatinib
  Other Names: Giotrif
Radiation: 2 Gy targeted radiotherapy
  Arms: Arm 2: Afatinib RP2D + 2 Gy targeted radiotherapy
Radiation: 4 Gy targeted radiotherapy
  Arms: Arm 3: Afatinib RP2D + 4 Gy targeted radiotherapy

SUMMARY:
Proof of principle phase 1b / randomised phase 2 study of afatinib penetration into cerebral metastases for patients undergoing neurosurgical resection, both with and without prior low-dose, targeted radiotherapy.

DETAILED DESCRIPTION:
Brain metastases occur in 20-40% of all patients with cancer, with an incidence 10 times higher than that of primary malignant brain tumours. patients with brain metastases are an underserved population. Overall they have a poor prognosis with a median survival of 1-2 months with corticosteroids and only 5-7 months after whole brain radiotherapy. An important factor in the poor prognosis of patients with brain metastases is the inability of many drugs to penetrate the blood-brain-barrier into tumour tissue.Combination therapy with surgical excision, radiotherapy and novel drugs could potentially improve the prognosis for some patients.

CamBMT1 is an open label, 3 Arm randomised Phase 2 trial investigating whether administration of a low dose of targeted radiotherapy during afatinib treatment could increase the concentration of drug penetration into brain metastases.

Eligible patients in Phase 2 will be randomised to 1 of 3 Arms:

Arm 1: no radiotherapy Arm 2: 2Gy radiotherapy Arm 3: 4Gy radiotherapy All patients will also receive 11 days of afatinib treatment at the recommended Phase 2 dose, previously determined in a Phase 1b safety run-in phase.

On Day 10, of afatinib treatment patients randomised to Arms 2 or 3 will receive their allocated dose of radiotherapy On Day 12, patients will undergo neurosurgical resection of their brain metastasis/ses.

Patients will be followed up on Day 22-28 and on Day 41 +/- 7 days

For the primary outcome measure, samples for measurement of plasma concentration of afatinib will be taken pre-treatment, on day 10 and Day 12 post-resection. Tumour tissue from the resected brain metastasis will be taken on day 12 for measurement of afatinib concentration. The primary outcome measure is the ratio of these concentrations.

The patient population studied will be breast/likely breast or lung/likely lung primary cancers with operable brain metastases.

ELIGIBILITY:
Inclusion Criteria

* Operable brain metastases from likely breast or lung origin as determined by local MDT. Both of the following groups of patients may be considered eligible:

  1. Patients with a past history of histologically/cytologically confirmed breast or lung cancer, now presenting with a new likely brain metastasis from that primary.
  2. Patients presenting with new, primary (breast/lung) tumours, plus synchronous, operable brain metastases, without pre-op tissue diagnosis.
* ECOG performance score 0, 1 or 2.
* Aged 18 years or older.
* Written informed consent.
* Patients are allowed to take oral corticosteroids however the plan should be for them to receive a stable dose of corticosteroids for at least 3 days before neurosurgery (i.e. trial days 10, 11, 12)

Exclusion Criteria

The presence of any of the following will preclude patient inclusion:

* History or presence of existing interstitial lung disease.
* Current clinically significant impairment of cardiac function (greater than Class II according to New York Heart Association [NYHA] classification).
* Unstable ischemic heart disease within the last 6 months, including myocardial infarction.
* Presence of QTc interval prolongation >480 ms.
* Clinically significant corneal or conjunctival eye disease.
* Clinically significant skin diseases such as psoriasis, rash or atopic dermatitis.
* Clinically significant impairment of GI function or GI disease including total gastrectomy that may alter the absorption of afatinib.
* Clinically significant, active peptic ulcer disease.
* Known positive test for human immunodeficiency virus (HIV), hepatitis B surface antigen (HBsAg) or hepatitis C virus (HCV) antibody or patients with any untreated serious infections.
* Pregnancy and contraception:

Female patients of child bearing potential must have a negative serum or urine pregnancy test within 14 days prior to registration/randomisation, and must use an effective method of contraception at least 1 week prior to treatment, during treatment and for at least 28 days after the final dose of study drug. Acceptable methods are:

True abstinence (this must be the patients usual and preferred lifestyle, not just for the duration of the study) Oral contraceptive (either combined or progestogen alone) Contraceptive implant, injections or patches Vaginal ring Intrauterine device (IUD, coil or intrauterine system) Condom and cap Diaphragm plus spermicide Tubal Ligation

* A female patient of child bearing potential is defined as a sexually mature woman not surgically sterilized or not post-menopausal for at least 24 consecutive months if aged 55 years or younger or 12 months if aged 56 years or older.
* Men must use one of the following, reliable forms to contraception for the entire duration of treatment and for 28 days after the final dose of study drug:

Condom plus spermicide even if female partner is using another method of contraception (Men should also use a condom to protect male partners, or female partners who are pregnant or breast feeding, from exposure to the study medicine in semen).

True abstinence (this must be the patients usual and preferred lifestyle, not just for the duration of the study)

* Concurrent severe and/or uncontrolled medical conditions (due to concurrent disease other than cancer) which in the opinion of the investigator could compromise participation in the study.
* Known or suspected active drug or alcohol abuse.
* Administration of chemotherapy, immunotherapy, radiotherapy or any investigational cancer therapy within 5 half-lives of the prior therapy or 2 weeks of first dose of afatinib, whichever is longer. Continuation of established endocrine therapy is allowed and no washout period is required. Established endocrine therapy (which may include GnRH analogues) is that which has been administered for at least 2 weeks prior to starting afatinib on Day 1
* Known hypersensitivity to afatinib or its excipients.
* Toxicities of prior therapies that have not resolved to ≤CTCAE Grade 1.
* Any of the following laboratory test findings:

Haemoglobin <90 g/L Absolute neutrophil count <1 x 109 /L Platelet count <100 x 109 /L AST or ALT >2.5 x upper limit of normal range (ULN) Total serum bilirubin >1.5 x ULN Creatinine >1.5 x ULN Creatinine clearance <30mL/min (Cockcroft-Gault)

* Patients taking potent P-gp inducers/inhibitors (see section 15.9)
* Any other reason which, in the opinion of the Investigator, interferes with the ability of the patient to participate in the study.
* Patients unable to comply with the protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2015-03-10 (Actual); Primary Completion 2020-08-12 (Actual); Study Completion 2021-08-12 (Actual)

PRIMARY OUTCOMES:
Ratio of afatinib concentration in: [resected brain metastases] / [plasma] - each measured in (ng/mL) on day 12 | Day 12 of treatment

SECONDARY OUTCOMES:
Safety of afatinib alone and combined with targeted low-dose radiotherapy - assessed by number of participants with treatment- related adverse events as assessed by CTCAE v4.0 | From consent to Day 41+/-7 days

CONTACTS AND LOCATIONS:
Overall Officials: Richard Baird, MD PhD, Principal Investigator — Cambridge University Hospitals NHS Foundation Trust
Locations (6):
- United Kingdom (6):
  - Cambridge University Hospitals NHS Foundation Trust, Cambridge, England
  - University Hospitals Birmingham NHS Foundation Trust, Birmingham
  - The Beatson West of Scotland Cancer Centre, Glasgow
  - Clatterbridge Cancer Centre, Liverpool
  - The Christie NHS Foundation Trust, Manchester
  - Oxford University Hospitals NHS Foundation Trust, Oxford